CLINICAL TRIAL: NCT03339635
Title: Short-term Testosterone Replacement in Testicular Cancer Survivors to Treat Overweight and Improve Cardiometabolic Risk: A Pilot Study
Brief Title: Short-term Testosterone Replacement in Testicular Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201600107
Record Dates: First submitted 2016-05-10; First posted 2017-11-13 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Testicular Cancer
MeSH Terms: conditions — Testicular Neoplasms | interventions — Testosterone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Testosterone gel (Experimental): Patients will be randomized to treatment with transdermal testosterone gel (Androgel) once daily during 20 weeks, followed by 20 weeks of active Androgel treatment in all participants.
  Interventions: Drug: Androgel (Testosterone gel)
- Placebo gel (Placebo Comparator): Patients will be randomized to treatment with placebo gel once daily during 20 weeks, followed by 20 weeks of active Androgel treatment in all participants.
  Interventions: Drug: Androgel (Testosterone gel); Drug: Placebo gel

INTERVENTIONS:
Drug: Androgel (Testosterone gel) — Patients will be randomized to treatment with transdermal testosterone gel (Androgel) once daily during 20 weeks, followed by 20 weeks of active Androgel treatment in all participants.
  Other Names: Androgel
Drug: Placebo gel — Patients will be randomized to treatment with transdermal placebo gel once daily during 20 weeks, followed by 20 weeks of active Androgel treatment in all participants.
  Other Names: Placebo
  Arms: Placebo gel

SUMMARY:
To assess the effects of testosterone replacement therapy on fat mass and other components of the metabolic syndrome. A randomized double-blind placebo controlled intervention study, followed by an open-label treatment phase. Results of this pilot study will be used to design a multicenter randomized controlled study in a large group of TC survivors

DETAILED DESCRIPTION:
Rationale: Testicular cancer (TC) survivors have an increased risk of hypogonadism (decreased testosterone and/or increased luteinizing hormone levels) and cardiovascular disease (CVD). Metabolic syndrome develops early after chemotherapy in 20-30% of long-term TC survivors and is associated with an increased risk of atherosclerotic disease in the general population. TC survivors who develop the metabolic syndrome have a higher body mass index (BMI) pretreatment, a larger BMI increase during follow-up, and lower total testosterone levels than patients without the metabolic syndrome. Testosterone replacement therapy as a short-term intervention during a limited time period may be an important strategy to reduce body weight and fat mass, restore cardiometabolic balance, and decrease the prevalence of the metabolic syndrome in TC survivors.

Objective: to assess the effects of testosterone replacement therapy on fat mass and other components of the metabolic syndrome.

Study design: randomized double-blind placebo controlled intervention study, followed by an open-label treatment phase. Results of this pilot study will be used to design a multicenter randomized controlled study in a large group of TC survivors

Study population: 40 TC patients, aged 18-55 years, at least 12 months after completion of curative treatment with unilateral orchidectomy and platinum-based chemotherapy, and having a fasting total testosterone level ≤12 nmol/l and a BMI ≥25 kg/m2.

Intervention: Patients will be randomized to treatment with transdermal testosterone gel (Androgel) or placebo gel once daily during 20 weeks, followed by 20 weeks of active Androgel treatment in all participants. The treatment dose will be 50 mg daily, adjusted to 25 mg in case of increased testosterone concentrations (average of 2 measurements >25 nmol/L) or signs of overdosing. Patients will be stratified according to testosterone level (8-12 nmol/L versus <8 nmol/L) and BMI (25-30 kg/m2 versus 30-35 kg/m2).

Main study parameters/endpoints: Primary endpoint is the change in fat mass as measured by Dual-Energy X-ray Absorption (DEXA) scan after 20 weeks of Androgel compared to placebo. Secondary endpoints are changes in fat mass between 20 and 40 weeks, and changes in abdominal visceral fat, BMI, adipocytokines, metabolic syndrome parameters, bone mass density, semen quality, sexual function, and quality of life between Androgel and placebo-treated patients.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study will provide an answer to the question whether testosterone replacement therapy as a short-term intervention has significant effects on obesity and fat metabolism and may, thus, reduce the prevalence of the metabolic syndrome in this population of young men with excellent long-term cancer-related prognosis, but an increased CVD risk. At various time points during the intervention, patients will be subjected to history taking and physical examination. Furthermore, blood will be drawn to: measure hormone levels, adipocytokines, lipids, glucose, insulin, and bone markers; to extract DNA for determination of gene polymorphisms; and to measure hematocrit and PSA as safety parameters. Semen analysis and a full body DEXA scan will be performed at 0, 20 and 40 weeks only. Patients will be asked to fill out questionnaires regarding quality of life, sexual health, and androgen deficiency symptoms at various time points during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with metastatic testicular cancer after unilateral orchidectomy and chemotherapy, at least 12 months after completion of last treatment and without evidence of disease. Combination chemotherapy should have contained a platinum compound, either cisplatin or carboplatin. In TC survivors, testosterone levels are routinely measured in blood during follow-up once every two years.
* Patients are eligible for screening if they are between 18 and 55 years of age
* have a documented low or low-normal total testosterone level ≤14 nmol/L, as measured during any of the follow-up visits, irrespective of signs and symptoms of androgen deficiency.

Eligible for actual study participation and randomization between Androgel and placebo will be:

* survivors of TC not using testosterone supplements, having biochemical evidence of hypogonadism (defined as a serum total testosterone concentration ≤ 12 nmol/L (345 ng/dL) measured after an overnight fast between 8:00 and 10:00 AM), and being overweight (as defined by a BMI ≥ 25 and <35 kg/m2).
* Patients should be able to understand and abide to the study protocol and sign written informed consent.

Exclusion Criteria:

* patients with a history of extragonadal testicular cancer
* patients planning to father children within the next 12 months
* patients taking corticosteroids or hormone replacement other than testosterone within 3 months of randomization
* patients taking medication with any antiandrogenic effects (e.g. spironolactone)
* patients with signs or history of hormone-dependent cancer (prostate or breast cancer)
* patients with severe lower urinary tract symptoms (as defined by International Prostate Symptom Score >19)
* patients with a history of coronary artery disease (angina pectoris, myocardial infarction) or heart failure
* patients with hematocrit >50%
* patients with untreated severe obstructive sleep apnea
* patients with uncontrolled hypertension
* patients with a BMI > 35 kg/m2
* patients with a history of epilepsy
* patients with debilitating psychiatric illness or inability to understand the study protocol, according to the opinion of the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
percent change in fat mass as measured using using full body dual X-ray absorptiometry | 20 weeks of treatment
  To assess the effects of 20 weeks of treatment with testosterone gel on fat mass as measured using full body dual X-ray absorptiometry (DEXA scan).

SECONDARY OUTCOMES:
Effect of treatment with testosterone gel | 20 and 40 weeks of treatment
  To assess the effects of 20 and 40 weeks of treatment with testosterone gel on obesity
Effect of treatment with testosterone gel | 20 and 40 weeks of treatment
  To assess the effects of 20 and 40 weeks of treatment with testosterone gel on signs and symptoms of hypogonadism

CONTACTS AND LOCATIONS:
Overall Officials: Janine Nuver, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No